CLINICAL TRIAL: NCT01318447
Title: International, Phase II Study of CyberKnife® for Hepatic Metastases From Colorectal Cancer
Brief Title: CyberKnife® for Hepatic Metastases From Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Accuray Incorporated (Industry)
Collaborators: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACC-HM-001
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Liver Metastases
Keywords: Hepatic metastases; Liver metastases; Colorectal cancer; Colorectal adenocarcinoma; Accuray; CyberKnife
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyberKnife SBRT (Experimental)
  Interventions: Radiation: CyberKnife SBRT

INTERVENTIONS:
Radiation: CyberKnife SBRT — Dose is 45 Gy (15 Gy in 3 fractions) and delivered over 5 to 10 days.

SUMMARY:
This prospective, multicenter study is intended to establish the efficacy and toxicity of treating unresectable colorectal liver metastases with accurately administered radiation using the CyberKnife stereotactic radiosurgery system.

DETAILED DESCRIPTION:
Colorectal cancer is the fourth most commonly diagnosed malignant disease worldwide, with an estimated 1,023,000 new cases and 529,000 deaths each year. The liver is the most frequent site of metastatic spread from colorectal cancer, 25% of colorectal cancer patients will have liver metastases at the time of initial colorectal resection and more than 50% of colorectal cancer patients will develop liver metastases during the course of the disease.

The current standard of care and only potential curative therapy for colorectal liver metastases is liver resection of the metastatic lesions. Surgical resection provides long term survival in patients with colorectal carcinoma (CRC) liver metastases. In a report of 1001 patients with metastatic colorectal cancer from Memorial Sloan-Kettering Cancer Center in NY, USA, surgical resection of liver metastases resulted in 3- and 5-year survival rates of 37% and 22%, respectively. Advances in pre- and intra-operative imaging and chemotherapy during recent years have increased overall survival up to 60% at 5 years after liver resection. However, 80-90% of liver metastases are unresectable at the time of diagnosis usually due to tumor location, multifocality, inadequate functional hepatic reserve or the patient's overall condition. For those patients, harboring unresectable liver metastases, alternative treatment approaches include neoadjuvant chemotherapy, local ablation therapy and stereotactic radiation therapy.

The recent availability of neoadjuvant chemotherapeutic agents has increased the response rates and doubled the median overall survival time for metastatic colorectal cancer from 10 to 20 months. Recent studies have demonstrated that neoadjuvant therapy allows 12.5% of patients with unresectable CRC liver metastases to be significantly downstaged and eligible for hepatic resection.

For unresectable CRC liver metastases, local ablative therapies are widely applied. Local ablative treatment refers to a variety of intervention techniques that specifically target tumors to directly destroy them. Numerous methods of ablation have been developed including cryoablation, percutaneous ethanol injection, radiofrequency ablation (RFA) and stereotactic radiation therapy. The most widely employed non-radiation based local ablative treatment is RFA which induces thermal ablation by passing high-frequency alternating current through the tumor utilizing electrodes that are placed within the tumor and surrounding tissue. RFA can be applied percutaneously under ultrasonic guidance or directly during laparoscopy or open laparotomy. Local recurrence rates of 44.4% at 18 months were reported by Solbiati et al. for CRC liver metastases with a median diameter of 2.6 cm. For tumors greater than 4 cm the local recurrence rate was 68%. RFA has an overall 3-year survival rate of 28-46% and a 5-year survival rate of 25%. However, patients with advanced hepatic decompensation, large tumors (3 to 5 cm), or multifocal tumors are generally considered poor candidates for RFA.

Conventional radiation therapy has been shown useful for palliation of hepatic capsular pain, but historically it has played a minor role in the treatment of patients with unresectable liver metastases. This can be attributed chiefly to the low tolerance of the whole liver to radiation. The liver was thought to be a relatively radiosensitive organ and with whole liver irradiation, it was difficult to achieve the radiation doses necessary to eradicate gross tumors without causing radiation induced liver disease. Partial liver irradiation has shown some promise. Limiting irradiation to only one-third of the liver through three-dimensional (3D) conformal radiotherapy techniques, including intensity modulated radiotherapy (IMRT), several studies have shown that partial liver irradiation is safe with doses up to 50-72.6 Gy. However, further dose escalation with conventional radiation therapy techniques risks injury to adjacent abdominal organs.

Stereotactic Body Radiation Therapy (SBRT) has emerged as a novel approach for the local ablation of liver metastases. SBRT provides a conformal isodose distribution with a steep radiation dose gradient allowing much higher doses of radiation than conventional radiation therapy and conformal radiotherapy techniques to be delivered safely with high precision to focal liver metastases while minimizing the radiation dose to normal liver and adjacent organs. To achieve this, precise localization of the target during treatment is required which necessitates accounting for tumor motion. SBRT technology utilizes a number of techniques to accommodate for tumor and respiratory motion including motion-restrictive techniques such as frames and abdominal compression, as well as motion-compensating techniques such as active breathing control and tumor tracking. The motion-restrictive techniques can be difficult for some patients to withstand, limiting those patients from being able to receive treatment. The motion-restrictive techniques can also necessitate the use of wide margins. Rusthoven et al. found a gross tumor volume (GTV) to planning target volume (PTV) expansion of up to 15 mm necessary in the craniocaudal direction. Wide margins can result in irradiation of a substantial volume of normal liver, potentially increasing the risk of radiation-induced injury. Some studies suggest the motion-compensating approach of active breathing control can aid in reducing the margins required by motion-restrictive approaches, however, Korreman et al. suggest those reductions may only be applicable with the use of image-guidance between and within sessions.

The CyberKnife robotic radiosurgery system (Accuray Incorporated, Sunnyvale, CA) an advanced platform to deliver SBRT, provides a therapeutic solution to this problem by continuously tracking the tumor during treatment while it accounts for organ motion due to respiratory movement, using the Synchrony respiratory tracking system (Accuray Incorporated, Sunnyvale, CA). Utilizing continuous tumor tracking, margin expansion to account for motion uncertainty can be reduced, having the potential to make this a safe and effective treatment. The frameless nature of the CyberKnife and its continuous image guidance system eliminates the need of motion-restriction techniques increasing the comfort and availability of the treatment to patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Hepatic metastases from histologically confirmed colorectal adenocarcinoma
* 3 hepatic lesions or less present
* Cumulative size of hepatic lesions between 1 and 10 cm
* Treatment determined by the liver/GI tumor board or equivalent organization at the participating site
* Metastatic disease not amenable to surgery as assessed by the panel (including a surgeon) or patient who refuses surgery
* Patient must be able to undergo contrast enhanced CT for planning
* Age >= 18 years old
* Performance Status (ECOG) ≤ 2
* Minimum of 6 months between the initial diagnosis of the disease and the first hepatic metastasis
* Minimum of 4 weeks between prior chemotherapy or targeted therapy and the first CyberKnife session
* Total bilirubin ≤ 3 times the upper limit of normal, ASAT and ALAT ≤ 5 times the upper limit of normal
* Albumin >= 36 g/L and lymphocytes >= 700/mm3
* No contraindication to fiducials implantation, hemostasis problems shall be corrected before implantation
* Life expectancy >= 3 months
* Patient affiliated with a health insurance system. Applicable for French patients only.
* Patient having signed the informed consent

Exclusion Criteria:

* Prior abdominal radiation therapy
* Any evidence of visible intra-hepatic bile duct dilatation on pre-treatment images
* Extrahepatic metastases
* Current evidence of ascitis
* Renal insufficiency (creatinine clearance < 45 ml/min)
* Known allergy to gold
* Pregnant or lactating woman
* Prior history of other cancer except basocellular carcinoma and in situ cervix carcinoma
* Patient already enrolled in another therapeutic clinical trial
* Inability to comply with follow-up visits for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Local recurrence-free survival | 12 months
  Local hepatic control (non progression: complete response, partial response or stable disease) will be assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Local recurrence-free survival time is calculated as the time between the date of first treatment session and the date of the first local recurrence. Patients alive who never experienced local recurrence at the time of analysis are censored at the date of the last follow-up visit. Patients who die from causes other than local recurrence at the time of analysis are censored at the date of death.

SECONDARY OUTCOMES:
Recurrence-free survival | 3, 6, 9, 12, 18 and 24 months
  Recurrence-free survival time is calculated as the time between the date of first treatment session and the date of a local or distant recurrence or death from progression whichever comes first. Patients alive who never experienced recurrence at the time of analysis are censored at the date of the last follow-up visit. Patients who die from causes other than cancer are censored at the date of death.
Overall survival | 3, 6, 9, 12, 18 and 24 months
  Overall survival time is calculated as the time between the date of first treatment session and the date of death, whatever the cause. Patients alive at the time of analysis are censored at the date of the last follow-up visit.
Acute and long term toxicity | 3, 6, 9, 12, 18 and 24 months
  The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for toxicity assessment.
Quality of Life | 3, 6, 9, 12, 18 and 24 months
  * European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) measures the quality of life for patients with cancer (for all participating sites).
  * Quality of Life Questionnaire-Liver Metastases Colorectal (QLQ-LMC21) is a specific module developed by the EORTC for patients with colorectal liver metastases (for sites in the United Kingdom, The Netherlands, Germany, France, and Belgium (French speaking part)).
Correlation of response as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST) | 6, 18 and 24 months
  The PERCIST response criteria will be applied to patients who have tumor characteristics measured by a PET-Scan. The association of response according to RECIST 1.1 and PERCIST will be evaluated with Spearman's correlation coefficient and the kappa statistic.
Local recurrence-free survival | 3, 6, 9, 18 and 24 months
  Local hepatic control (non progression: complete response, partial response or stable disease) will be assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Local recurrence-free survival time is calculated as the time between the date of first treatment session and the date of the first local recurrence. Patients alive who never experienced local recurrence at the time of analysis are censored at the date of the last follow-up visit. Patients who die from causes other than local recurrence at the time of analysis are censored at the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mirabel, MD, Principal Investigator — Centre Oscar Lambret
Locations (6):
- France (4):
  - Centre Antoine Lacassagne, Nice, France
  - Centre Oscar Lambret, Lille
  - Alexis Vautrin Cancer Center, Nancy
  - Hopital Bretonneau, Tours
- CyberKnife Zentrum Mecklenburg-Vorpommern, Güstrow, Germany, Germany
- Harley Street Clinic, London, United Kingdom